CLINICAL TRIAL: NCT03272152
Title: Comprehensive DNA Methylation Profiling of Inflammatory and Non-Inflammatory Mucosa in Crohn's Disease
Brief Title: Comprehensive DNA Methylation Profiling in Crohn's Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Jianan Ren, Director of General Surgery Institute, Jinling Hospital, China
Other Study IDs: 20170808
Record Dates: First submitted 2017-08-31; First posted 2017-09-05 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: Crohn Disease; Methylation; Illumina Human Methylation 850k BeadChip
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — inflamed and non-inflamed ileal mucosa of patients with Crohn's disease and normal ileal mucosa of healthy controls
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Inflamed CD group: Inflamed ileal mucosa was obtained from inflammed lesions of active CD patients
  Interventions: Genetic: Genome-wide DNA methylation
- Non-inflamed CD group: Non-inflamed ileal mucosa was obtained from normal sites of active CD patients
  Interventions: Genetic: Genome-wide DNA methylation
- Control group: Control ileal mucosa was obtained from healthy patients
  Interventions: Genetic: Genome-wide DNA methylation

INTERVENTIONS:
Genetic: Genome-wide DNA methylation — Genome-wide DNA methylation was determined using the Infinium Human Methylation 850K BeadChip.

SUMMARY:
Previous studies have indicated that abnormal DNA methylation frequently occurs in the mucosa in Crohn's disease. Comprehensive DNA methylation profiling of the inflamed and non-inflamed ileal mucosa of patients with Crohn's disease was performed. Genome-wide DNA methylation was determined using the Illumina HumanMethylation 850k BeadChip.

ELIGIBILITY:
Inclusion Criteria:

* Active Crohn's disease(CDAI score≥ 150)

Exclusion Criteria:

* No ileal lesions
* Under treatment of immunomodulators, biologic agents or steroids

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with active Crohn's disease who underwent colonoscopy at Jinling Hospital
Sampling Method: Non-Probability Sample
Enrollment: 14 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-09-30 (Estimated); Study Completion 2017-09-30 (Estimated)

PRIMARY OUTCOMES:
Intestinal inflammation under colonoscopy | Jan 2017 to Sep 2017
  Intestinal ulcer or enteritisis observed under colonoscopy

SECONDARY OUTCOMES:
CDAI | Jan 2017 to Sep 2017
  Crohns Disease Activity Index is measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Jinling Hospital, Nanjing, Jiangsu, China